CLINICAL TRIAL: NCT05438342
Title: An Expanded Clinical Study of Triple Therapy for Refractory Solid Tumors That Failed First-line Treatment for Recurrence and Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-IIT-021-E02
Record Dates: First submitted 2022-06-16; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- synchronized hyperthermia autologous progenitor expansion -T (SHAPE-T) (Experimental): Besides NCCN guideline recommended systemic anti-cancer treatment( chemotherapy /anti-PD-1 immmunotherapy/targeted therapy), combined with autoimmune cell therapy combined and noninvasive electromagnetic wave hyperthermia
  Interventions: Biological: Autologous Adoptive immune cells; Device: Thermotron RF-8EX; Drug: Chemotherapy，checkpoint immunotherapy, targeted therapy
- systemic anti-cancer treatment plus Hyperthermia (Active Comparator): BesidesNCCN guideline recommended systemic anti-cancer treatment( chemotherapy /anti-PD-1 immmunotherapy/targeted therapy), combined with noninvasive electromagnetic wave hyperthermia
  Interventions: Device: Thermotron RF-8EX; Drug: Chemotherapy，checkpoint immunotherapy, targeted therapy
- systemic anti-cancer treatment (Active Comparator): Only apply NCCN guideline recommended systemic anti-cancer treatment ( chemotherapy /anti-PD-1 immmunotherapy/targeted therapy)
  Interventions: Drug: Chemotherapy，checkpoint immunotherapy, targeted therapy

INTERVENTIONS:
Biological: Autologous Adoptive immune cells — Immunotherapy Mononuclear cells were collected from 50ml peripheral blood , and cultured adoptive immune cells for 15-20 days. Cells were infused back to the patients in 3 times via intravenous infusion.
  Arms: synchronized hyperthermia autologous progenitor expansion -T (SHAPE-T)
Device: Thermotron RF-8EX — Hyperthermia for 40-50 minutes
  Arms: synchronized hyperthermia autologous progenitor expansion -T (SHAPE-T); systemic anti-cancer treatment plus Hyperthermia
Drug: Chemotherapy，checkpoint immunotherapy, targeted therapy — The doctor chooses the appropriate systemic treatment for the patient based on NCCN guidelines

SUMMARY:
The clinical efficacy of chemotherapy /PD-1 monoclonal antibody/targeted therapy, chemotherapy /PD-1 monoclonal antibody/targeted therapy + noninvasive electromagnetic wave hyperthermia and chemotherapy /PD-1 monoclonal antibody/targeted therapy + noninvasive electromagnetic wave hyperthermia + autosomatic immunotherapy in the treatment of refractory refractory solid tumors with first-line treatment failure was compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously diagnosed with solid tumor by histopathology and/or cytology;
2. Aged 18 and 80, regardless of gender;
3. ECOG score of general physical condition was 0~2;
4. The expected survival time is at least 3 months;
5. Patients with metastatic and recurrent tumors who failed conventional first-line therapy (including those above first-line therapy) and need to change treatment regimens;
6. According to RECIST standards, at least one measurable objective tumor index (spiral CT detection target lesion 10mm);
7. WBC 3.0109 /L Hb 90g/L PLT 75.109 /L at baseline upon enrollment;
8. Normal liver function a) Liver: total bilirubin 2.0 mg/dL(34.2umol/L), 2.5 times the upper limit of AST and ALT, 5 times the upper limit of AST and ALT in patients with liver metastasis b) Kidney: Creatinine 2.5 mg/dL(221umol/L), creatinine clearance rate 60 mL/min;
9. Understand and sign informed consent and voluntarily participate in clinical research

Exclusion Criteria:

1. severe active infection and other serious complications;
2. Patients with a history of autoimmune diseases, including but not limited to multiple sclerosis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, excluding vitiligo;
3. Prednisone can be used in patients with systemic corticosteroid or other immunosuppressive hormone therapy. 0.5 mg/kg/day (maximum cell count group 40 mg/day) or other similar drugs in the same cell count group, inhaled corticosteroids for chronic obstructive pulmonary disease (COPD) or topical administration;
4. patients who have undergone major organ transplants;
5. Patients in the active stage of viral hepatitis;
6. Patients with coagulation dysfunction;
7. have uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia;
8. Pregnant or lactating women.
9. symptomatic brain metastases or mental disorders;
10. Participated in clinical trials of new drugs within 4 weeks before enrollment;
11. If the patients are randomly assigned to the hyperthermia treatment group, they need to refer to the exclusion requirements of hyperthermia (the hyperthermia site contains metal or thermal implant, skin allergy to heat, and body position cannot cooperate).
12. Other factors considered by researchers are not suitable for candidates.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  Frome the starting date of the enrollment until the date of the first documented disease progression or the date of the death from any cause,whichever comes first

SECONDARY OUTCOMES:
Overal survival(OS) | 24 months
  Frome the starting date of the enrollment until the date of the death from any cause
Safty(adverse events) | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Patient-Reported Outcome (PRO) | 24 months
  To assess and compare the PRO scores by patients in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ren, MD,PhD, Study Chair — Fudan University Pudong Medical Center
Locations (1):
- Fudan University Pudong Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No